CLINICAL TRIAL: NCT00060671
Title: An Open-Label, Randomized, Phase III Comparative Trial of BBR 2778 + Rituximab Versus Rituximab in the Treatment of Patients With Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma (NHL)
Brief Title: Comparative Trial for Pixantrone in Combination With Rituximab in Indolent Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZA III 02; NCT00062361 (obsolete NCT alias)
Record Dates: First submitted 2003-05-09; First posted 2003-05-12 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2013-05

CONDITIONS: Lymphoma, Follicular; Lymphoma, Mixed-Cell, Follicular; Lymphoma, Small Cleaved-Cell, Follicular; Lymphoma, Low-Grade
Keywords: Pixantrone; BBR 2778; chemotherapy; DNA Intercalator; Anthracycline; Rituximab; Rituxan; Mabthera; monoclonal antibody; antibody; NHL; Non-Hodgkin's lymphoma; indolent; low grade; Novuspharma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — Rituximab; pixantrone

INTERVENTIONS:
Drug: rituximab
Drug: Pixantrone (BBR 2778)

SUMMARY:
The purpose of this study is to determine whether combining pixantrone (BBR 2778, INN name pending) with the monoclonal antibody rituximab, leads to an increase in the period of patients' remission, compared to rituximab alone.

DETAILED DESCRIPTION:
This trial is being conducted in patients with indolent (or low-grade) non-Hodgkin's lymphoma, who have either relapsed or been refractory to previous treatment.

Pixantrone belongs to the DNA intercalator family of chemotherapy agents, which includes anthracyclines. DNA intercalators are commonly used to treat patients with indolent NHL, often in combination with the monoclonal antibody rituximab. This study represents the first large-scale, comparative trial in indolent NHL, designed to determine whether the response rate and time to tumour progression in patients treated with a combination of rituximab and a DNA intercalator, is significantly higher than seen in patients treated with rituximab alone.

This trial is randomized and controlled, which means that participating patients will be randomly assigned to one of two treatment groups:

1. Patients treated with both pixantrone and rituximab, in combination
2. Patients treated with only rituximab

This trial is expected to recruit around 800 patients in the US, Europe and Israel, with 400 patients recruited to each group.

Patients will be treated for around 18 weeks and will recieve regular physician monitoring for five years from the end of treatment.

ELIGIBILITY:
Inclusion criteria:

* Patients with relapsed or refractory indolent non-Hodgkin's lymphoma (NHL), including follicular lymphoma grade I and II
* Presenting with an episode of progressive disease, following 1-5 prior treatments (with either radiation, chemotherapy or rituximab).

Exclusion criteria:

* Patients that failed to respond to previous rituximab treatment, or relapsed within 6 months of the first rituximab infusion
* Patients known to have an allergic reaction to rituximab or murine derived proteins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2005-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Compare the time to tumor progression (TTP) of the combination of BBR 2778 (pixantrone) + rituximab with that of rituximab alone | For 5 years post treatment

SECONDARY OUTCOMES:
To compare BBR 2778 + rituximab versus rituximab for: | For 5 years post treatment
  * objective overall response rate (ORR; CR + PR)
  * objective complete response rate (CRR)
  * rate of molecular remission
  * time to response
  * time to complete response
  * duration of response
  * Time to Tumor Progression requiring treatment
  * Quality-Adjusted Time To Progression (QATTP)
  * overall survival
  * disease-specific survival
  * safety/tolerability

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Kenmar Research Institute, Los Angeles, California
  - Rocky Moutain Cancer Center, Denver, Colorado
  - Pasco, Hernando Oncology Associates, P.A., New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Orange Park Cancer Center, Orange Park, Florida
  - University of Chicago Medical Center Hematology / Oncology, Chicago, Illinois
  - Illinois Masonic Cancer Center, Chicago, Illinois
  - Edward Cancer Center, Naperville, Illinois
  - Hope Center, Terre Haute, Indiana
  - Commonwealth Hematology/Oncology, Danville, Kentucky
  - New England Hematology / Oncology Associates, Wellesley, Massachusetts
  - St. Joseph Oncology, Saint Joseph, Missouri
  - Christian Hospital, St Louis, Missouri
  - St. Johns Mercy Medical Center, St Louis, Missouri
  - Hematology - Oncology Centers of N. Rockies, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - East Orange VA Medical Center, East Orange, New Jersey
  - Hematology Oncology Associates of NJ, Paramus, New Jersey
  - Summit Medical Group/Overlook Onc Center, Summit, New Jersey
  - New Mexico Oncology / Hematology, Albuquerque, New Mexico
  - HemOnCare, P.C., Brooklyn, New York
  - Glens Falls Cancer Center, Glens Falls, New York
  - North Shore - Long Island Jewish Health System, New Hyde Park, New York
  - New York University, New York, New York
  - Upstate NY Cancer Research, Rochester, New York
  - South Shore Hematology-Oncology Associates, Rockville Centre, New York
  - Clinworks, Inc, Charlotte, North Carolina
  - Private Practice, Canton, Ohio
  - Blair Medical Associates, Altoona, Pennsylvania
  - Lancaster Cancer Center, LTD, Lancaster, Pennsylvania
  - Santee Hematology Oncology, Sumter, South Carolina
  - The West Clinic, Memphis, Tennessee
  - Central Utah Medical Clinic Hematology-Oncology, Provo, Utah
  - Oncology of Wisconsin, Glendale, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Rhinelander Regional Medical Group Onc., Rhinelander, Wisconsin

REFERENCES:
- [Result] Santoro A; Voglova J; Gabrail N; Ciuleanu T; Liberati M; Hancock BW; Stromatt S; Caballero D; Comparative Trial of Pixantrone + Rituximab vs Single agent Rituximab in the Treatment of Relapsed/Refractory Indolent Non-Hodgkin's Lymphoma; American Society of Clinical Oncology abstract and poster; Part 1, Vol 24 No 18S, June 20 supplement, 2006: 7578